CLINICAL TRIAL: NCT00565903
Title: Elucidating the Genetic Basis of the Pleuropulmonary Blastoma (PPB) Familial Cancer Syndrome
Acronym: PPB
Status: Completed | Type: Observational
Sponsor: Ashley Hill (Other)
Responsible Party: Sponsor-Investigator, Ashley Hill, MD, Professor of Pathology, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Other Study IDs: 05-0192 / 201012830
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Pleuropulmonary Blastoma; Cystic Nephroma; Sertoli-Leydig Cell Tumor of Ovary; Medulloepithelioma; Embryonal Rhabdomyosarcoma of Cervix; Goiter; Sarcoma; Pineoblastoma; Pituitary Tumors; Wilms Tumor
Keywords: pleuropulmonary blastoma; PPB; cystic nephroma; DICER1; miRNA
MeSH Terms: conditions — Pleuropulmonary blastoma; Sertoli-Leydig Cell Tumor; Neuroectodermal Tumors, Primitive; Goiter; Sarcoma; Pinealoma; Pituitary Neoplasms; Wilms Tumor

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We are collecting blood samples or saliva samples. When available, we also collect tumor samples from prior surgical procedures.
Oversight: Data Monitoring Committee: No

SUMMARY:
Pleuropulmonary Blastoma (PPB) is a rare lung tumor which develops in childhood. The underlying genetic factors which contribute to the development and progression of PPB are not defined. We are working to identify the genetic factors which may contribute to the development of this rare tumor.

DETAILED DESCRIPTION:
Studies of inherited cancer syndromes have provided unique opportunities to uncover and explain important cellular pathways with broad relevance to both sporadic cancers and human development. This proposal studies the cancer predisposition syndrome originally described as a familial form of pleuropulmonary blastoma (PPB). PPB is a rare, aggressive lung cancer that affects young children. Children with PPB and/or their family members are at increased risk for a number of rare conditions, including Wilms tumor, rhabdomyosarcoma, brain tumors, ovarian tumors and nodular hyperplasia of the thyroid gland. In 2009, we mapped a PPB locus and identified germline, loss of function mutations in one copy of DICER1 as the genetic basis of this syndrome. DICER1 encodes a protein that performs the final critical step in maturation of microRNAs (miRNAs). miRNAs are an important form of gene regulation. The syndrome's varied nature is likely attributable to the various roles of miRNAs during different developmental and/or functional circumstances. This study focuses on defining the full phenotype of this cancer predisposition syndrome including penetrance, expressivity in children and adults, pathologic classification of disease and spectrum of predisposing DICER1 mutations. Improved understanding of the clinical and genetic features of this cancer predisposition syndrome is essential to facilitate early diagnosis when the diseases are most curable, and to create genetic counseling and educational materials to guide medical care.

ELIGIBILITY:
Inclusion Criteria:

* Child or adult diagnosed with pleuropulmonary blastoma, cystic nephroma, embryonal rhabdomyosarcoma of uterine cervix, ovarian Sertoli-Leydig tumor or gynandroblastoma, pineoblastoma, pituitary blastoma, nasal chondromesenchymal hamartoma, medulloepithelioma, Wilms tumor, germline or mosaic DICER1 mutation

Exclusion Criteria:

* child or adult who does not fit inclusion criteria as listed above

Ages: 1 Day to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Families who have a child or adult with pleuropulmonary blastoma or cystic nephroma are invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 1247 (Actual)
Dates: Start 2005-03; Primary Completion 2018-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Identify the genetic factors which contribute to the development or progression of pleuropulmonary blastoma | 10 years

SECONDARY OUTCOMES:
Define the clinical features of the pleuropulmonary blastoma (PPB) familial cancer syndrome. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: D. Ashley Hill, MD, Study Chair — Children's National Research Institute; Kris Ann Schultz, MD, Study Director — Children's Hospital and Clinics of Minnesota
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
Sequence data deposited in ClinVar upon publication. Publication of all final results in NIHMS

REFERENCES:
- [Result] Schultz KAP, Williams GM, Kamihara J, Stewart DR, Harris AK, Bauer AJ, Turner J, Shah R, Schneider K, Schneider KW, Carr AG, Harney LA, Baldinger S, Frazier AL, Orbach D, Schneider DT, Malkin D, Dehner LP, Messinger YH, Hill DA. DICER1 and Associated Conditions: Identification of At-risk Individuals and Recommended Surveillance Strategies. Clin Cancer Res. 2018 May 15;24(10):2251-2261. doi: 10.1158/1078-0432.CCR-17-3089. Epub 2018 Jan 17. PMID 29343557
- [Result] Schultz KAP, Harris AK, Finch M, Dehner LP, Brown JB, Gershenson DM, Young RH, Field A, Yu W, Turner J, Cost NG, Schneider DT, Stewart DR, Frazier AL, Messinger Y, Hill DA. DICER1-related Sertoli-Leydig cell tumor and gynandroblastoma: Clinical and genetic findings from the International Ovarian and Testicular Stromal Tumor Registry. Gynecol Oncol. 2017 Dec;147(3):521-527. doi: 10.1016/j.ygyno.2017.09.034. Epub 2017 Oct 14. PMID 29037807
- [Result] Hill DA, Ivanovich J, Priest JR, Gurnett CA, Dehner LP, Desruisseau D, Jarzembowski JA, Wikenheiser-Brokamp KA, Suarez BK, Whelan AJ, Williams G, Bracamontes D, Messinger Y, Goodfellow PJ. DICER1 mutations in familial pleuropulmonary blastoma. Science. 2009 Aug 21;325(5943):965. doi: 10.1126/science.1174334. Epub 2009 Jun 25. PMID 19556464
- [Result] Pugh TJ, Yu W, Yang J, Field AL, Ambrogio L, Carter SL, Cibulskis K, Giannikopoulos P, Kiezun A, Kim J, McKenna A, Nickerson E, Getz G, Hoffher S, Messinger YH, Dehner LP, Roberts CW, Rodriguez-Galindo C, Williams GM, Rossi CT, Meyerson M, Hill DA. Exome sequencing of pleuropulmonary blastoma reveals frequent biallelic loss of TP53 and two hits in DICER1 resulting in retention of 5p-derived miRNA hairpin loop sequences. Oncogene. 2014 Nov 6;33(45):5295-302. doi: 10.1038/onc.2014.150. Epub 2014 Jun 9. PMID 24909177
- [Result] Schultz KA, Harris A, Williams GM, Baldinger S, Doros L, Valusek P, Frazier AL, Dehner LP, Messinger Y, Hill DA. Judicious DICER1 testing and surveillance imaging facilitates early diagnosis and cure of pleuropulmonary blastoma. Pediatr Blood Cancer. 2014 Sep;61(9):1695-7. doi: 10.1002/pbc.25092. Epub 2014 May 13. PMID 24821309
- [Result] Doros LA, Rossi CT, Yang J, Field A, Williams GM, Messinger Y, Cajaiba MM, Perlman EJ, A Schultz K, Cathro HP, Legallo RD, LaFortune KA, Chikwava KR, Faria P, Geller JI, Dome JS, Mullen EA, Gratias EJ, Dehner LP, Hill DA. DICER1 mutations in childhood cystic nephroma and its relationship to DICER1-renal sarcoma. Mod Pathol. 2014 Sep;27(9):1267-80. doi: 10.1038/modpathol.2013.242. Epub 2014 Jan 31. PMID 24481001
- [Result] Stewart DR, Messinger Y, Williams GM, Yang J, Field A, Schultz KA, Harney LA, Doros LA, Dehner LP, Hill DA. Nasal chondromesenchymal hamartomas arise secondary to germline and somatic mutations of DICER1 in the pleuropulmonary blastoma tumor predisposition disorder. Hum Genet. 2014 Nov;133(11):1443-50. doi: 10.1007/s00439-014-1474-9. Epub 2014 Aug 14. PMID 25118636
- [Result] Schultz KA, Yang J, Doros L, Williams GM, Harris A, Stewart DR, Messinger Y, Field A, Dehner LP, Hill DA. DICER1-pleuropulmonary blastoma familial tumor predisposition syndrome: a unique constellation of neoplastic conditions. Pathol Case Rev. 2014 Mar;19(2):90-100. doi: 10.1097/PCR.0000000000000027. PMID 25356068
- [Result] Messinger YH, Stewart DR, Priest JR, Williams GM, Harris AK, Schultz KA, Yang J, Doros L, Rosenberg PS, Hill DA, Dehner LP. Pleuropulmonary blastoma: a report on 350 central pathology-confirmed pleuropulmonary blastoma cases by the International Pleuropulmonary Blastoma Registry. Cancer. 2015 Jan 15;121(2):276-85. doi: 10.1002/cncr.29032. Epub 2014 Sep 10. PMID 25209242
- [Result] Rutter MM, Jha P, Schultz KA, Sheil A, Harris AK, Bauer AJ, Field AL, Geller J, Hill DA. DICER1 Mutations and Differentiated Thyroid Carcinoma: Evidence of a Direct Association. J Clin Endocrinol Metab. 2016 Jan;101(1):1-5. doi: 10.1210/jc.2015-2169. Epub 2015 Nov 10. PMID 26555935
- [Result] Khan NE, Bauer AJ, Schultz KAP, Doros L, Decastro RM, Ling A, Lodish MB, Harney LA, Kase RG, Carr AG, Rossi CT, Field A, Harris AK, Williams GM, Dehner LP, Messinger YH, Hill DA, Stewart DR. Quantification of Thyroid Cancer and Multinodular Goiter Risk in the DICER1 Syndrome: A Family-Based Cohort Study. J Clin Endocrinol Metab. 2017 May 1;102(5):1614-1622. doi: 10.1210/jc.2016-2954. PMID 28323992
- [Result] Kim J, Field A, Schultz KAP, Hill DA, Stewart DR. The prevalence of DICER1 pathogenic variation in population databases. Int J Cancer. 2017 Nov 15;141(10):2030-2036. doi: 10.1002/ijc.30907. Epub 2017 Aug 21. PMID 28748527
- [Result] Schultz KAP, Stewart DR, Kamihara J, Bauer AJ, Merideth MA, Stratton P, Huryn LA, Harris AK, Doros L, Field A, Carr AG, Dehner LP, Messinger Y, Hill DA. DICER1 Tumor Predisposition. 2014 Apr 24 [updated 2020 Apr 30]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK196157/ PMID 24761742
- [Result] Brenneman M, Field A, Yang J, Williams G, Doros L, Rossi C, Schultz KA, Rosenberg A, Ivanovich J, Turner J, Gordish-Dressman H, Stewart D, Yu W, Harris A, Schoettler P, Goodfellow P, Dehner L, Messinger Y, Hill DA. Temporal order of RNase IIIb and loss-of-function mutations during development determines phenotype in pleuropulmonary blastoma / DICER1 syndrome: a unique variant of the two-hit tumor suppression model. F1000Res. 2015 Jul 10;4:214. doi: 10.12688/f1000research.6746.2. eCollection 2015. PMID 26925222
- See also: PPB Research Program website — http://www.ppbgeneticstudy.org